CLINICAL TRIAL: NCT04315454
Title: The Analgesic Efficacy of Erector -Spinae Technique With Levobupvicaine in Patients Undergoing Upper Abdominal Cancer Surgery
Brief Title: Aalgesic Efficacy of Erector -Spinae Technique With Levobupvicaine in Patients Undergoing Upper Abdominal Cancer Surgery
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, Romany Gamal Rezk Bakeet, anesthesia specialist, South Egypt Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: southECI-1
Record Dates: First submitted 2020-03-13; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Erector Spinae Block Analgesia
MeSH Terms: interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Placebo Comparator): patients will receive 20 ml of normal saline into interfascial plane between rhomboids major &erector spinae muscle bilaterally at level thoracic spine T7,10 ml each side.
  Interventions: Drug: Levobupivacaine
- Group B (Experimental): Patients will receive 20 mg 0.25% Levobupivacaine into the interfascial plane between rhomboids major &erector spinae muscle bilaterally at level thoracic spine T7,10 ml each side.
  Interventions: Drug: Levobupivacaine

INTERVENTIONS:
Drug: Levobupivacaine — A group of patients will receive 20 ml of normal saline into the interfascial plane between rhomboids major &erector spinae muscle bilaterally at level thoracic spine T7,10 ml each side, the other group of patients will receive 20 mg 0.25% Levobupivacaine bilaterally as above 10 mg each side.

SUMMARY:
To study analgesic efficacy &safety of bilateral erector spinae block for upper abdominal cancer surgery as apart of multimodal analgesia.

DETAILED DESCRIPTION:
Patients will be randomly assigned using computer generated randomization program (http://www.randomizer.org) into two groups, each group of the them consist of 15 patients:

GROUP (A): {CONTROL GROUP} Patient will receive 20 ml of normal saline into interfascial plane between rhomboidus major &erector spinae muscle bilaterally at level thoracic spine T7,10 ml each side .

Group (B):

Patient will receive 20 mg 0.25% Levobupivacaine bilaterally as above 10 mg each side.

Preoperatively & post-operatively procedures:

Premedication will be given after complete fasting hours &after applying standard monitors (non invasive blood pressure, pulse oximetery, ECG, temperature and capnography, an intra-venous 16 gauge cannula will be inserted and secured).

Ultrasound guided Erector spinae plane block with patient in the sitting position & skin of the upper back is prepared with 2% chlorhexidine solution. Counting down from c7,the spine of T7 is identified it is corresponding to the tip the scapular spine ,a high frequency ultrasound probe is placed across T7 spine then probe move slowly laterally to identify transverse process of T7 ,So probe is moved to a vertical alignment and erector spinae muscle is visualized lying underneath the trapezius muscle.

Needle gauge will be inserted then 10 ml Levobupivacaine into interfascial plane between rhomboid major & erector spinae muscle in each side.

General anesthesia will be induced with Fentanyl 0.5 μg/kg, Propofol 2mg/kg, muscle relaxant (Atracurium 0.5 mg /kg) , inhalational anesthesia ( Isoflurane 1-1.5 MAC-or-sevoflurane2-3MAC ) as maintenance of anesthesia with frequent muscle relaxant every 20 minutes to maintain heart rate (HR) and blood pressure within 20% of the basal value. Patients were mechanically ventilated to maintain end tidal (ETCO2) between 35-40 mmHg. The inspired oxygen fraction (FIO2) was 0.5 using oxygen-and-air mixtures with frequent monitoring intraoperatively every 30 minutes, IV fentanyl infusion at rate of 0.1 μg/kg/hr may be used if needed.

Non steroidal anti-inflammatory as ketobrufen will be given intraoperatively at dose of (0.5-0.75mg/kg)then postoperatively every eight hours at the same dose.

The reverse of muscle relaxant with safe extubation will be done at the end of surgery.

-PCA morphine 2mg within five minutes lock out interval will be given postoperatively when there is pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient subjected to major upper abdominal cancer surgery.
* The enrolled age will be from 18-70 years old.
* ASA: I-III, NYHA: I-III.

Exclusion Criteria:

* ASA & physical status (NYHA) > III.
* Pregnant women.
* Body mass index >40 kg/m2.
* Pre-operative opioid consumption.
* Contraindication or patient's refusal of the procedure.
* Un co-operative patient.
* Coagulopathy, skin infection, significant organ dysfunction or drug allergy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
morphine consumption | 24 hours
  Decrease morphine consumption.

SECONDARY OUTCOMES:
VAS score | 24 hours
  Intensity of pain at rest and during pain-provoking movements (deep breathing,coughing, mobilization) measured by VAS pain score immediately postoperative then at 2, 4 ,6 ,12& 24 hours after surgery}
patient satisfaction | 24 hours
  patient satisfaction in the first 24 hour post operatively.
Hemodynamic | 24 hours
  - Hemodynamic variables including (systolic and diastolic BP, heart rate, oxygen saturation & respiratory rate) measured preoperatively (baseline measurement) then immediately postoperative and at 2, 4 ,6 ,12& 24 hours after surgery.
blood gas | 24 hours
  -Blood gases will be drawn preoperatively and at 12 hour interval in the PACU for assessment of Oxygen tension (PO2) & Co2 tension (PCO2).

CONTACTS AND LOCATIONS:
Overall Officials: Romany G. Rezk, MSc, Principal Investigator — Specialist
Locations (1):
- South Egypt Cancer Institute, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
as we should ask patients and take their consents to share these date